CLINICAL TRIAL: NCT06869083
Title: Application-Delivered Patient Education in Enhancing the Usage of Apixaban in Patients With Atrial Fibrillation: Randomized Control Therapy
Brief Title: Application-Delivered Patient Education in Enhancing the Usage of Apixaban in Patients With Atrial Fibrillation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2024-1210
Record Dates: First submitted 2025-02-20; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation on Apixaban Treatment
Keywords: atrial fibrillation; apixaban; anticoagulation; adherence; application; eduction
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App education group (Experimental)
  Interventions: Other: AF application enhancing AF education and drug adhrence
- No-App education group (Active Comparator)
  Interventions: Other: AF application without enhancing AF education and drug adhrence

INTERVENTIONS:
Other: AF application enhancing AF education and drug adhrence — This group will use AF-application. The app will include content related to anticoagulation therapy, such as: medication reminders or intake confirmation for anticoagulants, the importance of anticoagulation therapy in stroke prevention, the role of antiarrhythmic and rate-control medications in symptom management, the necessity of controlling risk factors such as hypertension, diabetes, and hyperlipidemia, and quality of life and cognitive function assessments through questionnaires.
  Arms: App education group
Other: AF application without enhancing AF education and drug adhrence — This group will use AF-application. However, this application will not contain materials enhancing AF education and adherence.
  Arms: No-App education group

SUMMARY:
"AF is the most common arrhythmia, with an overall prevalence of approximately 2%. It is particularly prevalent in individuals over 60 years old, affecting about 5% of this population. With the aging population, the global prevalence of AF is increasing. In South Korea, the overall prevalence of AF increased from 0.73% in 2006 to 1.53% in 2015, a 2.1-fold increase. By 2060, it is projected that 2.3 million people in Korea will have AF, with a prevalence rate of 5.81%. AF accounts for approximately 20% of all ischemic strokes, and patients with AF have an annual risk of ischemic stroke ranging from 6% to 10%. Additionally, AF can lead to heart failure and doubles the mortality rate. Despite various treatment options, the mortality rate associated with AF continues to rise annually.

Anticoagulation therapy for the prevention of thromboembolism in AF is a crucial treatment approach. Traditional warfarin therapy has been shown to reduce the risk of stroke by approximately 63%. Recently developed non-vitamin K oral anticoagulants (NOACs) have demonstrated similar efficacy to warfarin while offering a lower risk of hemorrhagic complications, particularly intracranial hemorrhage, making them a safer alternative.

Adherence to anticoagulant therapy is crucial for the effective prevention of stroke in patients with AF. Poor adherence to anticoagulants significantly increases the risk of thromboembolic events, including ischemic stroke. Studies have shown that patients with low adherence to anticoagulation therapy experience higher rates of stroke and mortality compared to those who consistently take their medication as prescribed. Ensuring proper adherence to anticoagulants, whether traditional warfarin or newer non-vitamin K oral anticoagulants (NOACs), is essential to maximizing treatment benefits while minimizing complications. Factors influencing adherence include medication side effects, complexity of the treatment regimen, patient awareness, and regular follow-up with healthcare providers. Strategies to improve adherence, such as patient education, simplified dosing regimens, and routine monitoring, play a key role in reducing the burden of AF-related strokes.

The burden of cardiovascular risk factors, including lifestyle factors and borderline conditions, as well as comorbidities, significantly influences both the risk of AF development and its prognosis. The continuum of unhealthy lifestyle habits, risk factors, and cardiovascular diseases contributes to atrial remodeling, cardiomyopathy, and ultimately, the onset of AF through the combined effects of multiple interacting factors. One of the three core components of the Atrial Fibrillation Better Care (ABC) pathway for comprehensive AF management is the ""C"" component, which focuses on the identification and management of comorbidities, cardiometabolic risk factors, and unhealthy lifestyle habits. Effective management of these risk factors and cardiovascular diseases plays a crucial role in stroke prevention and in reducing AF burden and symptom severity. Recent randomized clinical trials have shown that targeted treatment of underlying conditions improves the maintenance of sinus rhythm following AF ablation in patients with persistent AF and heart failure.

Education by healthcare providers regarding medication adherence and risk factor management for existing AF patients is often limited due to constraints in manpower and resources. However, leveraging new technologies such as mobile applications can help overcome these limitations by enhancing patient education and improving medication adherence without the need for additional healthcare personnel.

This study is fundamentally a prospective, multicenter, randomized, open-label clinical trial. Patients with atrial fibrillation who are prescribed edoxaban at participating institutions will be randomly assigned to either an app-based anticoagulation education group or a non-education group. Primary objective is to demonstrate that an app-based education program for patients with AF taking apixaban results in a lower incidence of major cardiovascular events (ischemic stroke/systemic embolism, major bleeding, hospitalization, myocardial infarction, and death) compared to the non-education group. Secondary Objective is to investigate the impact of the intervention on secondary events, including stroke, systemic embolism, transient ischemic attack (TIA), major bleeding, non-major bleeding, hospitalization, myocardial infarction, death, and medication adherence. Exploratory Objective are to assess treatment satisfaction using the Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) questionnaire, and to evaluate cognitive function changes using the Korean Dementia Screening Questionnaire (KDSQ).

DETAILED DESCRIPTION:
"This study is fundamentally a prospective, multicenter, randomized, open-label clinical trial. Patients with AF receiving apixaban at participating institutions will be randomly assigned to either an app-based anticoagulation education group or a non-education group. The incidence rates of primary, secondary, and exploratory events will be assessed.

The app will include content related to anticoagulation therapy, such as: medication reminders or intake confirmation for anticoagulants, the importance of anticoagulation therapy in stroke prevention, the role of antiarrhythmic and rate-control medications in symptom management, the necessity of controlling risk factors such as hypertension, diabetes, and hyperlipidemia, and quality of life and cognitive function assessments through questionnaires.

Follow-up assessments will be conducted every six months after enrollment. The anticipated enrollment period is four years, with a minimum follow-up duration of one year.

Participants will have voluntary access to educational materials in the app. Medication adherence will be encouraged through reminder alarms, while other educational components will not have specific evaluation methods. The study investigator is responsible for developing the medication adherence education app. The app's content is currently being finalized, and development will be completed using research funding after study approval.

Randomization will be conducted using an Excel macro function, assigning participants in a 1:1 ratio. The randomization process will be uploaded to iCReaT, an electronic case report form (eCRF) system, allowing verification at the time of participant registration.

Primary Outcome: The primary composite outcome consists of ischemic stroke, intracranial hemorrhage, and myocardial infarction. This outcome was selected based on previous domestic studies demonstrating that medication adherence reduces the incidence of these composite events. Evaluations will be conducted every six months after enrollment. The anticipated enrollment period is four years, with a minimum follow-up duration of one year.

Secondary Outcomes: The study will assess the following secondary outcomes: Stroke (ischemic and hemorrhagic), Transient ischemic attack (TIA), Systemic embolism, Major bleeding, Non-major bleeding, Myocardial infarction, Death, Hospitalization events, and Medication adherence. Evaluations will be conducted every six months after enrollment. The anticipated enrollment period is four years, with a minimum follow-up duration of one year.

"

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older with non-valvular atrial fibrillation (NVAF).
* Willingness to provide informed consent and participate in the study.
* Receiving Elxaban as anticoagulation therapy.
* Ability to use the mobile application.

Exclusion Criteria:

* Inability to understand the study or refusal to provide consent.
* Minors under 19 years of age.
* Pregnant or breastfeeding women.
* Conditions requiring chronic anticoagulation therapy other than atrial fibrillation (e.g., mechanical heart valve replacement).
* Life expectancy of less than one year due to severe comorbid conditions.
* Contraindications to Elxaban use, including:

  1. Hypersensitivity to the active ingredient or any excipients of the drug.
  2. Severe renal impairment (CrCL <15 mL/min).
  3. Clinically significant active bleeding.
  4. Increased bleeding risk due to the following conditions:

     * Recent history of gastrointestinal ulcer.
     * High-risk malignant neoplasms.
     * Recent brain or spinal cord injury.
     * Recent history of brain, spinal, or ophthalmic surgery.
     * Recent history of intracranial or cerebral hemorrhage.
     * Suspected or confirmed esophageal varices.
     * Arteriovenous malformations.
     * Vascular aneurysms.
     * Spinal or intracranial vascular abnormalities.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5200 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
The primary composite outcome | every 6 month up to 4 years until the end of study, with a minum follow-up duration of one year.
  The primary composite outcome consists of ischemic stroke, intracranial hemorrhage, and myocardial infarction.

SECONDARY OUTCOMES:
Secondary end points assessed time to stroke (ischemic and hemorrhagic) | every 6 month up to 4 years until the end of study
transient ischemic attack (TIA) | every 6 month up to 4 years until the end of study
systemic embolism | every 6 month up to 4 years until the end of study
major bleeding | every 6 month up to 4 years until the end of study
  Major bleeding was defined according to the criteria of International Society on Thrombosis and Haemostasis (ISTH).
clinically relevant non-major bleeding | every 6 month up to 4 years until the end of study
  Clinically relevant non-major bleeding define a bleeding event that is neither a major bleed as defined by the ISTH 1 nor a non-clinically consequential minor bleeding event.
myocardial infarction | every 6 month up to 4 years until the end of study
death | every 6 month up to 4 years until the end of study
hospitalization events | every 6 month up to 4 years until the end of study
medication adherence | every 6 month up to 4 years until the end of study
  Medication adherence is defined as the percentage of the prescribed doses of the medication actually taken by the patient over a follow-up duration.
Secondary end points assessed time to stroke (ischemic and hemorrhagic) | a minum follow-up duration of one year.
transient ischemic attack (TIA) | a minum follow-up duration of one year.
systemic embolism | a minum follow-up duration of one year.
major bleeding | a minum follow-up duration of one year.
  Major bleeding was defined according to the criteria of International Society on Thrombosis and Haemostasis (ISTH).
clinically relevant non-major bleeding | a minum follow-up duration of one year.
  Clinically relevant non-major bleeding define a bleeding event that is neither a major bleed as defined by the ISTH 1 nor a non-clinically consequential minor bleeding event.
myocardial infarction | a minum follow-up duration of one year.
death | a minum follow-up duration of one year.
hospitalization events | a minum follow-up duration of one year.
medication adherence | a minum follow-up duration of one year.
  Medication adherence is defined as the percentage of the prescribed doses of the medication actually taken by the patient over a follow-up duration.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided